CLINICAL TRIAL: NCT02740673
Title: Testing Cognitive Functions in Patients With COPD Using a Driving Simulator
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Driving simulator, COPD, v.2
Record Dates: First submitted 2015-12-28; First posted 2016-04-15 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Driving simulator (Other): Using the driving simulator for 30 min.
  Interventions: Device: Driving simulator

INTERVENTIONS:
Device: Driving simulator — Patients are asked to use a driving simulator to test their driving skills

SUMMARY:
Little is known about the causes and degree of cognitive dysfunction in patients with Chronic Obstructive Pulmonary Disease (COPD), especially their driving abilities. The purpose of the study is to examine the cognitive skills of patients with COPD by using a driving simulator and to examine correlations to factors that may predict cognitive dysfunction in these patients.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD (Forced Expiratory Volume in 1 second (FEV1) / Forced Vital Capacity (FVC) < 0,70)
* no exacerbations within the last 6 weeks
* valid driver's license and having driven a car within the last 3 months

Exclusion Criteria:

* lacking the ability to use the driving simulator
* no valid driver's license
* alcohol abuse (> 21 units per week)
* a known diagnosis of obstructive sleep apnea
* uncorrected impaired vision or hearing
* unstable ischemic heart disease, left-sided heart failure, severe neurologic diseases, cancer, severe peripheral vascular disease, severe psychiatric diseases, former apoplexia and uncontrolled hypertension, thyroid diseases or diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Standard deviation from the centre of the road | During the 30 min. of driving in the simulator
  Measuring how far from the centre of the road the patient has been driving in the driving simulation
Number of nil responses | During the 30 min. of driving in the simulator
  Measuring the number of times the patients doesn't react to the number "2" on the screen
Response time | During the 30 min. of driving in the simulator
  Measuring the mean amount of response time from the number "2" appears on the screen until the patient reacts
Number of off-road events per hour | During the 30 min. of driving in the simulator
  The number of times the car is off-road during the driving simulation

SECONDARY OUTCOMES:
Number of patients with comorbidities | At enrolment
  Patients with comorbidities will be registered
Lung function tests | At enrolment
Depression and anxiety | At enrolment
  Using the Hospital Anxiety and Depression Scale
Cognitive functions | At enrolment
  Using the Mini Mental State Examination and the Clock Drawing Test

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Prior, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark